CLINICAL TRIAL: NCT07322042
Title: Evaluating Screening Adherence Between Moment for Parents App and Attention Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poisera, Inc. (Industry)
Collaborators: University of Michigan (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: R43MH130293 (NIH); R43MH130293 (NIH)
Record Dates: First submitted 2025-12-08; First posted 2026-01-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Screening Adherence
Keywords: maternal mental health; perinatal mood and anxiety disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moment for Parents Intervention (Experimental): Participants in the intervention arm will use the full Moment for Parents mobile application, which includes an interactive chatbot that delivers brief lessons, mood check-ins, guided reflections, and optional mindfulness activities. Lessons are grouped into topic-based "Journeys," each consisting of short modules designed to support emotional well-being during pregnancy and postpartum. The app sends daily push notifications prompting users to continue their Journey or engage with mood-related activities. Standard mental health screening instruments (PHQ-9 and GAD-7) are integrated into these check-ins, allowing screening to occur naturally within regular app use. The intervention is designed to increase user engagement and create more opportunities for mental health screening completion than traditional perinatal care.
  Interventions: Behavioral: Perinatal Psychoeducation Articles; Behavioral: Bi-weekly Perinatal Mental Health Screening; Behavioral: Chatbot-Guided Journaling; Behavioral: Perinatal-Focused Meditations; Behavioral: Themed Perinatal Learning Pathways
- Moment for Parents Attention Control (Sham Comparator): Participants in the attention control arm will use a modified version of the Moment for Parents mobile application that does not include the interactive chatbot or guided "Journey" lessons. Instead, the app sends weekly push notifications prompting users to read brief educational articles on pregnancy and postpartum topics, including infant development and common maternal experiences. The app delivers the same mental health screeners (PHQ-9 and GAD-7) at comparable intervals as the intervention arm. However, the screeners are not embedded within conversational features. This version of the app provides exposure to perinatal health information without the personalized engagement strategies present in the intervention condition.
  Interventions: Behavioral: Perinatal Psychoeducation Articles; Behavioral: Bi-weekly Perinatal Mental Health Screening

INTERVENTIONS:
Behavioral: Perinatal Psychoeducation Articles — Participants access brief, evidence-based articles related to pregnancy, postpartum experiences, and infant development. Articles are designed to increase perinatal knowledge and normalize common emotional and physical changes during this period.
Behavioral: Bi-weekly Perinatal Mental Health Screening — Participants complete validated mental health screening tools (PHQ-9 and GAD-7) integrated into a mobile app. This allows screening to occur in a non-clinical, routine format and increases opportunities for early symptom identification.
Behavioral: Chatbot-Guided Journaling — Participants interact with a conversational chatbot that guides them through mood reflection prompts, journaling activities, and emotional processing exercises. The chatbot personalizes the experience using user input and delivers supportive, non-clinical language to reduce barriers to disclosure.
  Arms: Moment for Parents Intervention
Behavioral: Perinatal-Focused Meditations — Participants are provided optional audio-based mindfulness and self-regulation meditations tailored to pregnancy and postpartum stressors. These meditations support emotional regulation and help participants manage worry, fatigue, and distress.
  Arms: Moment for Parents Intervention
Behavioral: Themed Perinatal Learning Pathways — Participants select topic-based curricula (called "Journeys") composed of brief lessons that include educational content, reflections, and optional activities. Each pathway focuses on a specific aspect of pregnancy or postpartum well-being (e.g., resilience, social support, communication with clinicians) and prompts sustained engagement through short, sequential modules.
  Arms: Moment for Parents Intervention

SUMMARY:
Mental health challenges, such as depression and anxiety, are the most common medical complications during pregnancy and after childbirth. Many women experience these symptoms, yet half are never screened, let alone diagnosed. When mental health concerns go unnoticed, they can affect a mother's well-being, her birth experience, and her child's development. When identified early, these conditions are treatable. However, current healthcare practices often fail to screen women consistently, and many women do not feel comfortable discussing emotional struggles with healthcare providers.

This study will test whether a mobile app called Moment for Parents can help pregnant and postpartum women complete mental health screenings more regularly. The app includes educational articles, guided reflections, and mood check-ins that help women explore their feelings in a private, supportive environment. The app also includes a chatbot that guides them through short lessons about motherhood, stress, relationships, and emotional well-being. These conversations are designed to feel friendly and relatable, like talking with a knowledgeable companion rather than filling out a medical form. The investigators expect that this more personal experience may make it easier for women to notice and track changes in their mental health and encourage them to complete regular screeners.

The study will enroll 160 women who are pregnant or within the first year after giving birth. Participants will be randomly assigned to one of two groups:

Intervention group: Uses the full Moment for Parents app, including the interactive chatbot.

Control group: Uses a simplified version of the app with weekly articles but no chatbot.

Both groups will receive mental health screenings through the app over a 12-week period. These screenings include standard, widely used questionnaires that measure symptoms of depression and anxiety.

If a participant's answers show signs of concerning symptoms, such as depression, anxiety, or thoughts of self-harm, the study team will connect her to licensed mental health professionals for support. This offers more rapid help than the current standard of care, which often screens women only once during pregnancy.

The investigators hypothesize that women who interact with the chatbot version of the Moment for Parents app will complete mental health screenings twice as often as women using the app without the chatbot. In other words, the investigators believe the chatbot will increase regular screening by creating a more engaging and supportive experience.

Increasing the number of completed mental health screenings could help identify emotional struggles earlier, when treatment is most effective. If this study shows that the Moment for Parents app improves screening and engagement, it could guide the design of a larger study and help shape future care for pregnant and postpartum women nationwide. Overall, this research aims to make mental health support more accessible, less stigmatizing, and easier to use.

DETAILED DESCRIPTION:
This study is a 12-week, two-arm pilot randomized controlled trial (RCT) designed to evaluate whether an interactive mobile application, the Moment for Parents app, improves adherence to routine mental health screening among pregnant and postpartum women. Perinatal mood and anxiety disorders (PMADs) are prevalent, impactful on maternal and infant health, and often remain undetected due to stigma, inconsistent clinical screening practices, and limited engagement with healthcare systems. Digital screening embedded within a consumer-facing app may address these barriers by normalizing emotional check-ins, reducing self-presentation concerns, and enabling repeated screening opportunities over time.

Participants will be randomized 1:1 to either (1) the Moment for Parents chatbot intervention arm or (2) an attention control arm. Randomization will occur automatically at enrollment using permuted block randomization with a fixed block size to ensure balanced allocation across key baseline characteristics (e.g., race, gestational age, mental health history). Because all data are collected through the app platform, independent assessor blinding is not required.

The intervention arm receives the fully developed Moment for Parents application, which includes interactive chatbot-guided lessons, reflective prompts, mood check-ins, and optional audio-based meditations. These components are organized into topic-based "Journeys," each composed of short lessons designed to be completed in approximately five minutes. The chatbot integrates validated mental health screeners (PHQ-9 and GAD-7) within regular mood check-ins, allowing screening to be delivered contextually rather than as a standalone questionnaire. Participants receive daily push notifications encouraging continued engagement.

The control arm receives a modified version of the Moment for Parents app that omits the chatbot and interactive lesson structure. Instead, users receive weekly push notifications linking to educational articles describing expected changes during pregnancy and postpartum, including infant development and maternal physical and emotional adjustments. Like the intervention arm, mental health screening is administered via the app algorithm at regular intervals, ensuring both groups receive equivalent exposure to screening opportunities.

The primary focus of the trial is to compare screening adherence trajectories between arms. Both the timing and frequency of PHQ-9 and GAD-7 administration exceed current clinical norms, which typically involve only one screening during the perinatal period. Screening and engagement metrics are passively captured through the app backend, allowing complete ascertainment of screening adherence without missing data due to participant attrition.

Participants who exceed clinical cutoffs for depression, anxiety, or suicidality will be automatically flagged via an application programming interface (API) that alerts a licensed behavioral health team affiliated with the MC3 Perinatal Program. This clinical escalation pathway includes structured risk assessment and, when indicated, facilitated linkage to psychiatric care. These clinical procedures are not part of the research intervention itself and are governed by independent IRB oversight within the MC3 program.

In addition to comparing screening adherence between arms, the study will evaluate user engagement behaviors, identify participant-level predictors of engagement, and explore patterns of app utilization over time. Quantitative app usage data, such as screens completed, content viewed, and activities initiated, will be analyzed alongside qualitative interview data from participants demonstrating high product affinity. These findings will inform optimization of the intervention and guide sample stratification strategies for a future, fully powered Phase II randomized trial.

The proposed research aims to address a major gap in perinatal mental health care by testing whether a mobile behavioral health tool can feasibly support sustained screening adherence outside of clinical environments. If successful, this approach may enable earlier identification of PMAD symptoms, reduce disparities in detection and treatment, and provide empirical evidence supporting digital engagement pathways for perinatal mental health monitoring at scale.

ELIGIBILITY:
Inclusion Criteria:

Women who are:

* Pregnant or up to 1 year postpartum
* Age 18 years or older
* Lives in Michigan
* Owns a smartphone with internet access
* Proficient in English

Exclusion Criteria:

* Not female
* Not currently pregnant or more than 1 year postpartum
* Younger than 18 years old
* Does not live in Michigan
* Does not own a smartphone with internet access
* Not proficient in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mental Health Screening Adherence | From enrollment to 12 weeks post-enrollment
  Mental health screening adherence will be measured as the total number of completed PHQ-9 and GAD-7 screenings delivered through the Moment for Parents app during the 12-week study period. Screening opportunities occur bi-weekly and are recorded passively by the application backend, allowing precise tracking of whether a participant completed each scheduled screening. Adherence will be compared across study arms using count-based analysis methods to determine whether the interactive chatbot increases screening adherence relative to the attention control condition.

SECONDARY OUTCOMES:
App Engagement | From enrollment to 12 weeks post-enrollment
  Engagement will be measured using backend app analytics, including counts of completed chatbot conversations, articles read, meditations accessed, and activities saved. Engagement rate will be calculated as the average number of activities completed per active user within each weekly interval.
App Retention | From enrollment to 12 weeks post-enrollment
  App retention will be measured as the length of time a participant continues to actively engage with the Moment for Parents application from initial use until the final recorded activity (e.g., chatbot interaction, article read, or meditation completed). Retention patterns will be analyzed to determine how long participants remain active in the app environment and whether retention differs between study arms or varies by baseline characteristics such as mental health history or initial engagement levels.
Baseline Predictors of Screening Adherence | From enrollment to 12 weeks post-enrollment
  We will use Cox proportional hazards regression to examine predictors, including demographics, mental health history, and baseline PHQ-9 and GAD-7 score. As above, the starting point will be when the participant enrolls in the study and completes the first PHQ-9 and GAD-7 screen, and the endpoint will be when she completes her final PHQ-9 and GAD-7 screen. The proportional hazards assumption will be tested for each predictor by including the interaction between the predictor and time. If the interaction term is significant, we will include it in the final model to account for the non-proportional hazards. For each predictor, we will report the odds ratio with 95% CI.
Patterns of Mental Health Screening Behavior | From enrollment to 12 weeks post-enrollment
  Patterns of screening behavior will be evaluated by modeling the binary outcome of whether participants complete the PHQ-9 and GAD-7 screeners each week using a generalized linear mixed-effects model with a logit link. Graphical analyses of fitted model estimates over the 12-week period will be used to identify distinct user subgroups (e.g., "early adopters," "infrequent responders," and "compliers") based on trajectories of screening completion. Comparisons will be made between study arms and across participant characteristics (such as baseline mental health history and initial screening scores) to determine whether these factors are associated with differing patterns of screening behavior.
Perceived Value of the Moment for Parents App | From 1 week after enrollment through 12 weeks after enrollment
  Using a four-item product-market fit survey, participants will report perceived benefit, emotional response if access were removed, and suggested improvements. Responses from the "Very disappointed" subgroup will be used to identify the characteristics of users who perceive high value.
Thematic Insights from User Experience Interviews | From 1 week after enrollment through 3 months after enrollment
  Semi-structured interviews with participants who report being "very disappointed" at the prospect of losing access to the app will be analyzed using inductive thematic analysis to identify common needs, experiences, and features associated with meaningful engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Kerppola, MBA, MSc, Principal Investigator — Poisera, Inc.; Maria Muzik, MD, MSc, Principal Investigator — University of Michigan
Locations (1):
- Remote/Virtual Participation, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared in de-identified form for the primary and secondary outcome measures described in the study protocol. All identifiers (such as names, contact information, and geographic data that could permit re-identification) will be removed prior to sharing. De-identified datasets will include only outcome variables and relevant demographic variables needed for reproducibility.
  Data will be made available upon reasonable request to qualified researchers whose proposed use is consistent with the goals of the study and who agree to comply with data use and confidentiality requirements. Data will be provided after study completion and primary results publication. No identifiable information collected as part of the Moment for Parents platform or clinical escalation procedures will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified individual participant data and supporting documentation will be made available beginning 6 months after publication of the primary study results and will remain available for 3 years thereafter.
Access Criteria: Access will be granted to investigators affiliated with academic, nonprofit, or government research institutions who submit a methodologically sound request and sign a data use agreement outlining requirements for confidentiality and appropriate data handling.

REFERENCES:
- See also: Study Recruitment and Enrollment Information — https://www.momentforparents.com/research

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT07322042/Prot_SAP_000.pdf
  • Informed Consent Form (2026-02-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT07322042/ICF_002.pdf